CLINICAL TRIAL: NCT00989261
Title: Phase 2 Open-Label, AC220 Monotherapy Efficacy (ACE) Study in Patients With Acute Myeloid Leukemia (AML) With and Without FLT3-ITD Activating Mutations
Brief Title: Efficacy Study for AC220 to Treat Acute Myeloid Leukemia (AML)
Acronym: ACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-002; 2009-013093-41 (EudraCT Number)
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; AC220; acute; FLT3; inhibitor; kinase; leukemia; leukaemia; myeloid; relapsed; refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Recurrence | interventions — quizartinib; Powders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1; ≥60 years of age (Experimental): Participants ≥60 years of age who were relapsed after one first-line chemotherapy regimen (with or without consolidation) and after first complete remission <12 months or are primary refractory to first-line chemotherapy received a starting dose of 200 mg/day quizartinib.
  Exploratory: FLT3-ITD (+) and FLT3-ITD (-) Confirmatory: FLT3-ITD (+) and FLT3-ITD (-)
  After an amendment, male participants received a starting dose of 135 mg/day quizartinib and all females received a starting dose of 90 mg/day.
  Interventions: Drug: Compound AC220
- Cohort 2; ≥18 years of age (Experimental): Participants ≥18 years of age (including participants ≥60 years of age) who were relapsed or refractory after one second-line (salvage) regimen or after hematopoietic stem cell transplant (HSCT) received a starting dose of 200 mg/day quizartinib.
  Exploratory: FLT3-ITD (+) and FLT3-ITD (-) Confirmatory: FLT3-ITD (+) and FLT3-ITD (-)
  After an amendment, male participants received a starting dose of 135 mg/day quizartinib and all females received a starting dose of 90 mg/day.
  Interventions: Drug: Compound AC220

INTERVENTIONS:
Drug: Compound AC220 — Precomplexed powder in bottle formulation supplied as 200 mg in a 60 cc polyethylene terephthalate (PET) plastic bottle. Requires reconstitution by a pharmacist, must be stored securely, and protected from light.
  Other Names: AC010220 × 2HCl, oral powder for reconstitution

SUMMARY:
AC220 will be administered as a once daily oral solution given continuously as 28-day treatment cycles, without any rest periods, until disease progression, relapse, intolerance to the drug, or elective allogeneic hematopoietic stem cell transplantation (HSCT).

ELIGIBILITY:
Current enrollment is open only to FLT3-ITD positive, Cohort 1.

Inclusion Criteria:

1. Males and females age ≥18 years in second relapse or refractory.
2. Males and females age ≥60 years in first relapse or refractory.
3. Must have baseline bone marrow sample taken.
4. Morphologically documented primary AML or AML secondary to myelodysplastic syndrome (MDS with ≥20% bone marrow or peripheral blasts), as defined by the World Health Organization (WHO) criteria, confirmed by pathology review at treating institution.
5. Able to swallow the liquid study drug.
6. Eastern Cooperative Oncology Group performance status of 0 to 2
7. In the absence of rapidly progressing disease, the interval from prior treatment to time of AC220 administration will be at least 2 weeks for cytotoxic agents or at least 5 half-lives for noncytotoxic agents. The use of chemotherapeutic or antileukemic agents other than hydroxyurea is not permitted during the study with the possible exception of intrathecal (IT) therapy at the discretion of the Investigator and with the agreement of the Sponsor.
8. Persistent chronic clinically significant non-hematological toxicities from prior treatment must be ≤Grade 1.
9. Prior therapy with FLT3 inhibitors is permitted, except previous treatment with AC220.
10. Serum creatinine ≤1.5 × upper limit of normal (ULN) and glomerular filtration rate (GFR) > 30 mL/min
11. Serum potassium, magnesium, and calcium levels should be at least within institutional normal limits.
12. Total serum bilirubin ≤1.5 × ULN
13. Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤2.5 × ULN
14. Females of childbearing potential must have a negative pregnancy test (urine β-hCG).
15. Females of childbearing potential and sexually mature males must agree to use a medically accepted method of contraception throughout the study.
16. Written informed consent must be provided.

Exclusion Criteria:

1. Patients over the age of 85 years except at the discretion of the Investigator and with agreement of the Sponsor.
2. Diagnosis of acute promyelocytic leukemia
3. Diagnosis of chronic myelogenous leukemia (CML) in blast crisis
4. AML in relapse or refractory after 3 or more previous lines of chemotherapy (and/or HSCT) treatment
5. AML or antecedent MDS secondary to prior chemotherapy
6. Persistent clinically significant non-hematological toxicity that is Grade >1 by NCI CTCAE v4 from prior chemotherapy
7. Patients who have had HSCT and are within 100 days of transplant and/or are still taking immunosuppressive drugs and/or have clinically significant graft-versus-host disease requiring treatment and/or have >Grade 1 persistent non hematological toxicity related to the transplant
8. Clinically active central nervous system (CNS) leukemia. Patients with CNS leukemia, which is controlled, but who are still receiving IT therapy at study entry may be considered eligible and continue receive IT therapy at the discretion of the Investigator and with agreement of the Sponsor.
9. Patients who have previously received AC220
10. Disseminated intravascular coagulation (DIC) (diagnosis by laboratory or clinical assessment)
11. Major surgery within 4 weeks prior to enrollment in the study
12. Radiation therapy within 4 weeks prior to, or concurrent with study
13. Use of concomitant drugs that prolong the time between the start of the Q wave and the end of the T wave (QT)/corrected interval between the Q wave and T wave (QTc) interval and/or are CYP3A4 inhibitors are prohibited with the exception of antibiotics, antifungals, and other antimicrobials that are used as standard of care to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the patient.
14. Uncontrolled or significant cardiovascular disease
15. Women who are pregnant, lactating, or unwilling to use contraception if of childbearing potential
16. Men who are unwilling to use contraception if their partners are of childbearing potential
17. Active, uncontrolled infection
18. Human immunodeficiency virus positivity
19. Active hepatitis B or C or other active liver disease
20. History of cancer, except Stage 1 cervix or nonmelanotic skin cancer, with the possible exception of patients in complete remission

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09-28 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Interim Chief Medical Officer, Study Director — Ambit Biosciences Corporation
Locations (85):
- United States (20):
  - University of California, San Francisco, San Francisco, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Clinical Trials Center, Nashville, Tennessee
  - The Vanderbuilt Clinic, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (15):
  - Institut Paoli Calmettes Centre Regional de Lutte Contre le Cancer, Marseille, Cedex 9
  - Hematologie - CHU Purpan, Toulouse, Cedex
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Universitaire d'Angers, d'Angers
  - Centre Hospitalier Universitaire Grenoble, Grenoble
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire Limoges, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital Saint-Antoine, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - Centre Henry Becquerel, Service d'Hematologie, Rouen
  - Centre Hospitalier Regional Universitaire, Hopital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire Brabois, Vandœuvre-lès-Nancy
- Germany (21):
  - Charite Campus Virchow Klinikum, Berlin
  - Charite, Campus Benjamin Franklin, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Unikliniksklinikum Carl Gustav Carus, Dresden
  - Uniklinik Essen, Westdeutsches Tumorzentrum, Essen
  - Klinikum der Johann Wolfgang Goethe Universitat, Frankfurt am Main
  - Asklepios Klinik St Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Leipzig Selbstandige Abteilung fur Hamatologie, Leipzig
  - Universitatsklinikum Magdeburg, Magdeburg
  - Universitatsklinikum Mannheim, Mannheim
  - Philipps-Universitat Marburg, Marburg
  - Klinikum rechts der Isar, Technische Universitat Munchen, München
  - Universitatsklinikum Munster, Münster
  - Universitatsklinikum Regensburg Abteilung fur Hamatologie, Regensburg
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - Universitatsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (11):
  - Instituto Di Ematologia "L.Ea. Seragnoli", Bologna
  - Unita Trapianti di Midollo Osseo per Adulti, Brescia
  - Presidio Ospedaliero "A. Businco" - Centro di Riferimento Oncologico Regionale, Cagliari
  - Azienda Ospedaliera-Universitaria Vittorio Emanuele-Ferrarotto, Catania
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Farmacia Ospidaliera, Orbassano
  - Ospedale Civile S. Maria delle Croci, Ravenna
  - Ospedale Sant Eugenio, Roma
  - Universita Degli Studi di Roma Tor Vergata, Roma
  - Azienda Ospedaliero Universitaria Senese, Siena
  - Azienda Ospedaliero Universitaria S. Maria della Misericordia di Udine, Clinica Ematologica, Udine
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Utrecht University Medical Centre, Dept. of Hematology, Utrecht
- Dolnoslaskie Centrum Transplantacji Komorkowych z, Wroclaw, Poland
- Spain (9):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catala d'Oncologia del Hospital Universitari Germans, Barcelona
  - Instituto Catalan de Oncologia-Hospital Universitari de Girona, Girona
  - Hospital de la Princesa, Servicio de Hematologia, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario de Salamanca, Hospital Clinico, Servicio de Hematologia, Salamanca
  - Hospital La Fe, Servicio de Hematologia, Valencia
- United Kingdom (5):
  - Addenbrook's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Saint James University Hospital, Institute of Oncology, Leeds
  - Hanmmersmith Hospital, Dept. of Hematology, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Cortes J, Perl AE, Dohner H, Kantarjian H, Martinelli G, Kovacsovics T, Rousselot P, Steffen B, Dombret H, Estey E, Strickland S, Altman JK, Baldus CD, Burnett A, Kramer A, Russell N, Shah NP, Smith CC, Wang ES, Ifrah N, Gammon G, Trone D, Lazzaretto D, Levis M. Quizartinib, an FLT3 inhibitor, as monotherapy in patients with relapsed or refractory acute myeloid leukaemia: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2018 Jul;19(7):889-903. doi: 10.1016/S1470-2045(18)30240-7. Epub 2018 May 31. PMID 29859851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 333 participants from 9 countries (United States, Germany, France, Italy, United Kingdom, Spain, Netherlands, Canada, and Poland) who met all inclusion and none of the exclusion criteria were included in the study.
Pre-assignment Details: All participants in both cohorts initially received a starting dose of 200 mg/day quizartinib (maximum tolerated dose). To ensure complete inhibition of FLT3, all male subjects in both cohorts later received a starting dose of 135 mg/day quizartinib, and all females received a starting dose of 90 mg/day.
Period: Overall Study
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Started | 157 | 176
Completed | 142 | 154
Not Completed | 15 | 22
Not completed — Still in follow up | 12 | 21
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age | Total
Number analyzed (Participants) | 157 | 176 | 333
Age, Continuous [Median (Full Range); unit: years] | 69.0 [32 to 86] | 51.0 [19 to 77] | 63.0 [19 to 86]
Age, Customized [Count of Participants; unit: Participants]
  Less than 60 years | 2 | 132 | 134
  At least 60 years | 155 | 44 | 199
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 163
  Male | 77 | 93 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 126 | 150 | 276
  Unknown or Not Reported | 27 | 20 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 5 | 10
  White | 135 | 156 | 291
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 12 | 4 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 4
  Netherlands | 5 | 5 | 10
  United States | 59 | 86 | 145
  Poland | 2 | 0 | 2
  Italy | 16 | 12 | 28
  United Kingdom | 7 | 7 | 14
  France | 24 | 29 | 53
  Germany | 37 | 27 | 64
  Spain | 5 | 8 | 13
Weight [Mean (Standard Deviation); unit: kg] | 74.66 (14.75) | 74.76 (19.41) | 74.72 (17.33)

OUTCOME MEASURES:

1. Primary Outcome: Derived Disease Assessment Based on Local Morphology Including All On-Treatment Data (Safety Population, FLT3-ITD [+] Participants)
Description: Derived disease assessment based on local morphology of bone marrow disease performed by each local site pathologist, including all on-treatment data (Safety Population, FLT3-ITD[+] Participants)
  Modified from Cheson et al, abbreviations include the following: CR=complete remission; CRc=composite complete remission (CR+CRp+CRi); CRi=complete remission with incomplete hematological recovery, includes participants who met CRia criteria plus participants who met CRib criteria; CRia=all criteria specified for CR are met except for incomplete hematological recovery with residual neutropenia <1 x 10^9/L with or without complete platelet recovery. Red blood cell and platelet transfusion independence is not required; CRib=All criteria for CR or CRp are met, except for recent red blood cell or platelet transfusion; CRp=complete remission with incomplete platelet recovery; NR=no response; PR=partial remission.
Time Frame: Within the first 3 cycles of treatment (84 days)
Population: Derived disease assessments were conducted in the Safety Population (FLT3-ITD [+] participants).
Measure: Number; unit: participants
Groups:
- Cohort 1; ≥60 Years of Age: Participants ≥60 years of age who were relapsed after one first-line chemotherapy regimen (with or without consolidation) and after first complete remission <12 months or are primary refractory to first-line chemotherapy received a starting dose of 200 mg/day quizartinib.
  * Exploratory (N=24): FLT3-ITD(+): n=22; FLT3-ITD(-): n=2; unknown: n=0
  * Confirmatory (N=133): FLT3-ITD(+): n=90; FLT3-ITD(-): n=42; unknown: n=1
  * Total (N=157): FLT3-ITD (+): n=112; FLT3-ITD(-): n=44; unknown: n=1
  After an amendment, male participants received a starting dose of 135 mg/day quizartinib and all females received a starting dose of 90 mg/day.
- Cohort 2; ≥18 Years of Age: Participants ≥18 years of age (including participants ≥60 years of age) who were relapsed or refractory after one second-line (salvage) regimen or after hematopoietic stem cell transplant (HSCT) received a starting dose of 200 mg/day quizartinib.
  * Exploratory (N=38): FLT3-ITD(+): n=36; FLT3-ITD(-): n=2; unknown: n=0
  * Confirmatory (N=138): FLT3-ITD(+): n=100; FLT3-ITD(-): n=38; unknown: n=0
  Total (N=176): FLT3-ITD(+): n=136; FLT3-ITD(-): n=40; unknown: n=0
  After an amendment, male participants received a starting dose of 135 mg/day quizartinib and all females received a starting dose of 90 mg/day.
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 112 | 136
participants
  Composite complete remission (CRc) | 63 | 62
  Complete remission (CR) | 3 | 5
  Complete remission with incomplete platelet (CRp) | 4 | 2
  Complete remission with incomplete hematologic CRi | 56 | 55
  Partial remission (PR) | 23 | 39
  No response (NR) | 20 | 24
  Unknown | 6 | 11

2. Primary Outcome: Derived Disease Assessment Based on Local Morphology Including All On-Treatment Data (Safety Population, FLT3-ITD [-] Participants)
Description: Derived disease assessment based on local morphology of bone marrow disease performed by each local site pathologist, including all on-treatment data (Safety Population, FLT3-ITD[-] Participants)
  Modified from Cheson et al, abbreviations include the following: CR=complete remission; CRc=composite complete remission (CR+CRp+CRi); CRi=complete remission with incomplete hematological recovery, includes participants who met CRia criteria plus participants who met CRib criteria; CRia=all criteria specified for CR are met except for incomplete hematological recovery with residual neutropenia <1 x 10^9/L with or without complete platelet recovery. Red blood cell and platelet transfusion independence is not required; CRib=All criteria for CR or CRp are met, except for recent red blood cell or platelet transfusion; CRp=complete remission with incomplete platelet recovery; NR=no response; PR=partial remission.
Time Frame: Within the first 3 cycles of treatment (84 days)
Population: Derived disease assessments were conducted in the Safety Population (FLT3-ITD [-] participants).
Measure: Number; unit: participants
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 44 | 40
participants
  Composite complete remission (CRc) | 16 | 12
  Complete remission (CR) | 2 | 1
  Complete remission with incomplete platelet (CRp) | 1 | 1
  Complete remission with incomplete hematologic CRi | 13 | 10
  Partial remission (PR) | 4 | 6
  No response (NR) | 17 | 16
  Unknown | 7 | 6

3. Primary Outcome: Number of Participants With Composite Complete Remission (CRc), Categorised by FLT3-ITD Status
Description: CRc is defined as composite complete remission (CR+CRp+CRi) - CR = complete remission; CRp = complete remission with incomplete platelet recovery; CRi = complete remission with incomplete hematological recovery, includes participants who met CRia criteria plus participants who met CRib criteria; CRia = all criteria specified for CR are met except for incomplete hematological recovery with residual neutropenia <1 x 10^9/L with or without complete platelet recovery. Red blood cell and platelet transfusion independence is not required; CRib = all criteria for CR or CRp are met, except for recent red blood cell or platelet transfusion.
Time Frame: within 28 months
Population: Composite complete remission was assessed in the Safety Population.
Measure: Number; unit: participants
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 157 | 176
participants
  FLT3-ITD(+) | 63 | 62
  FLT3-ITD(-) | 16 | 12

4. Secondary Outcome: Duration of Composite Complete Remission in FLT3-ITD (+) Participants Who Achieved CRc Based on All On-Treatment Data
Description: Kaplan-Meier analysis of duration of composite complete remission derived based on local morphology including all on-treatment data (Safety Population).
  The definition of relapse at CRc includes an evaluation of blasts in the peripheral blood of >1%.Though not specified in the protocol, the addition of these criteria was deemed necessary for consistency with the Cheson criteria.
Time Frame: From time at which CRc was achieved until disease progression or death, up to approximately 3 years post treatment
Population: Duration of composite complete remission was assessed in the Safety Population based on FLT3-ITD (+) participants available for this analysis (Cohort 1: n=63; Cohort 2: n=62).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 63 | 62
weeks | 12.1 [6.3 to 15.7] | 10.6 [8.1 to 16.1]

5. Secondary Outcome: Duration of Composite Complete Remission in FLT3-ITD (-) Participants Who Achieved CRc Based on All On-Treatment Data
Description: as for outcome 4
Time Frame: From time at which CRc was achieved until disease progression or death, up to approximately 3 years post treatment
Population: Duration of composite complete remission was assessed in the Safety Population based on FLT3-ITD (-) participants available for this analysis (Cohort 1: n=16; Cohort 2: n=12).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 16 | 12
weeks | 16.4 [8.1 to 30.4] | 7.0 [4.1 to 8.1]

6. Secondary Outcome: Duration of Any Response in FLT3-ITD (+) Participants
Description: Kaplan-Meier analysis of duration of any response (CR, CRp, CRi, or PR), derived based on local morphology for participants who achieved a response during the first 3 cycles of treatment (Safety Population).
Time Frame: From the time of any response until disease progression or death, up to approximately 3 years post treatment
Population: Response (based on local morphology) was assessed in the Safety Population (FLT3-ITD [+] participants).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 83 | 99
weeks | 15.7 [14.1 to 21.3] | 14.1 [11.1 to 22.3]

7. Secondary Outcome: Duration of Any Response in FLT3-ITD (-) Participants
Description: as for outcome 6
Time Frame: From the time of any response until disease progression or death, up to approximately 3 years post treatment
Population: Response (based on local morphology) was assessed in the Safety Population (FLT3-ITD [-] participants).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 20 | 18
weeks | 22.4 [10.1 to 34.1] | 8.1 [7.4 to 8.1]

8. Secondary Outcome: Median Duration of Leukemia-free Survival in FLT3-ITD (+) Participants
Description: Kaplan-Meier analysis of leukemia-free survival in participants who achieved a CRc in the first three cycles of treatment derived based on local morphology (Safety Population).
Time Frame: From the time CRc was achieved until disease progression or death, up to approximately 3 years post treatment
Population: Leukemia-free survival (based on local morphology) was assessed in the Safety Population (FLT3-ITD [+] participants).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 61 | 61
weeks | 12.1 [6.1 to 14.3] | 12.9 [9.4 to 19.1]

9. Secondary Outcome: Median Duration of Leukemia-free Survival in FLT3-ITD (-) Participants
Description: as for outcome 8
Time Frame: From the time CRc was achieved until disease progression or death, up to approximately 3 years post treatment
Population: Leukemia-free survival (based on local morphology) was assessed in the Safety Population (FLT3-ITD [-] participants).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 14 | 11
weeks | 16.4 [8.1 to 26.1] | 7.0 [5.0 to 8.1]

10. Secondary Outcome: Median Duration of Overall Survival in FLT3-ITD (+) Participants
Description: Kaplan-Meier analysis of overall survival (Safety Population)
Time Frame: Time from first dose to death from any cause, up to 3 years post treatment
Population: Overall survival was assessed in the Safety Population (FLT3-ITD [+] participants).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 112 | 136
weeks | 25.4 [21.3 to 29.7] | 24.0 [21.1 to 27.1]

11. Secondary Outcome: Median Duration of Overall Survival in FLT3-ITD (-) Participants
Description: Kaplan-Meier analysis of overall survival (Safety Population)
Time Frame: Time from first dose to death from any cause, up to approximately 3 years post treatment
Population: Overall survival was assessed in the Safety Population (FLT3-ITD [-] participants).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 44 | 40
weeks | 19.1 [12.0 to 29.4] | 25.1 [18.1 to 37.0]

12. Secondary Outcome: Early Treatment-related Death
Description: Early treatment-related deaths included all treatment-related deaths prior to the end of Cycle 3 with a 3-day window (Cycle 3 end date + 3 days), unless the death was following a CRc response assessed by the Investigator.
Time Frame: Within first 3 cycles of treatment (84 days)
Population: Early treatment-related deaths were assessed in the Safety Population.
Measure: Number; unit: participants
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
Number analyzed (Participants) | 157 | 176
participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected after the first dose of study drug through 30 days after the last dose of study drug, approximately 5 years.
Description: Of note, AML disease progression (which includes the verbatim terms of progressive disease, disease progression, and relapsed AML) is reported as an AE in the data output and in the in-text tables; however, it is not considered an AE because of the population under study and is not further discussed.
Groups:
- Cohort 1; ≥60 Years of Age: FLT3-ITD positive and negative populations will be divided into 2 cohorts as follows:
  Participants ≥60 years of age who were relapsed after one first-line chemotherapy regimen (with or without consolidation) and after first complete remission <12 months or are primary refractory to first-line chemotherapy received a starting dose of 200 mg/day quizartinib.
  Exploratory: FLT3-ITD (+) and FLT3-ITD (-) Confirmatory: FLT3-ITD (+) and FLT3-ITD (-)
  After an amendment, male participants received a starting dose of 135 mg/day quizartinib and all females received a starting dose of 90 mg/day.
Arm/Group | Cohort 1; ≥60 Years of Age | Cohort 2; ≥18 Years of Age
All-Cause Mortality (participants affected / at risk) | 71/157 | 60/176
Serious Adverse Events (participants affected / at risk) | 134/157 | 135/176
Other Adverse Events (participants affected / at risk) | 151/157 | 175/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1; ≥60 Years of Age (N=157) | Cohort 2; ≥18 Years of Age (N=176)
Hematoma (Vascular disorders) | 1 | 3
Hemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 0
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 | 36
Leukemic infiltration brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphohistiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Graft versus host disease in skin (Immune system disorders) | 0 | 1
Asthenia (General disorders) | 2 | 1
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 2 | 4
Localized edema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 2
Edema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 10 | 8
Secretion discharge (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 3 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Accidental poisoning (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 3 | 0
Subdural hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 4
Blood potassium decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 17 | 16
Hepatic enzyme increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 3
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Acute promyelocytic leukemia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 7 | 6
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 60 | 66
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6
Aphasia (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Hemorrhage intracranial (Nervous system disorders) | 4 | 1
Hemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Intraventricular hemorrhage (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient ischemic attack (Nervous system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Barrett's esophagus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
Mouth hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Hematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 2
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Acinetobacter bacteremia (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1
Bacteremia (Infections and infestations) | 6 | 4
Bacterial sepsis (Infections and infestations) | 2 | 2
Breast cellulitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 1
Candidiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 5 | 3
Cellulitis orbital (Infections and infestations) | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 4
Enterobacter bacteremia (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 2
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia bacteremia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Gingival infection (Infections and infestations) | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Klebsiella bacteremia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 6
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 0
Necrotizing fascitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pericoronitis (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 24 | 16
Pneumonia fungal (Infections and infestations) | 1 | 7
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pseudomonal bacteremia (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection fungal (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 12 | 13
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 3 | 3
Serratia bacteremia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Sinusitis fungal (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal bacteremia (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 2 | 3
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 6
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1; ≥60 Years of Age (N=157) | Cohort 2; ≥18 Years of Age (N=176)
Hematoma (Vascular disorders) | 17 (17) | 12 (12)
Hypotension (Vascular disorders) | 17 (17) | 13 (13)
Asthenia (General disorders) | 33 (33) | 32 (32)
Chest pain (General disorders) | 10 (10) | 13 (13)
Chills (General disorders) | 13 (13) | 14 (14)
Fatigue (General disorders) | 62 (62) | 49 (49)
Mucosal inflammation (General disorders) | 8 (8) | 15 (15)
Edema peripheral (General disorders) | 46 (46) | 45 (45)
Pyrexia (General disorders) | 47 (47) | 49 (49)
Confusional state (Psychiatric disorders) | 8 (8) | 2 (2)
Depression (Psychiatric disorders) | 12 (12) | 10 (10)
Insomnia (Psychiatric disorders) | 11 (11) | 15 (15)
Contusion (Injury, poisoning and procedural complications) | 14 (14) | 6 (6)
Alanine aminotransferse increased (Investigations) | 9 (9) | 15 (15)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 7 (7)
Electrocardiogram QT prolonged (Investigations) | 31 (31) | 48 (48)
Neutrophil count decreased (Investigations) | 8 (8) | 6 (6)
Platelet count decreased (Investigations) | 17 (17) | 12 (12)
Weight decreased (Investigations) | 10 (10) | 11 (11)
Tachycardia (Cardiac disorders) | 10 (10) | 10 (10)
Anemia (Blood and lymphatic system disorders) | 44 (44) | 48 (48)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12) | 14 (14)
Leukopenia (Blood and lymphatic system disorders) | 10 (10) | 18 (18)
Neutropenia (Blood and lymphatic system disorders) | 15 (15) | 20 (20)
Pancytopenia (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (22) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 37 (37)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 26 (26)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 27 (27)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (12)
Dizziness (Nervous system disorders) | 27 (27) | 18 (18)
Dysgeusia (Nervous system disorders) | 44 (44) | 34 (34)
Headache (Nervous system disorders) | 19 (19) | 24 (24)
Paresthesia (Nervous system disorders) | 13 (13) | 5 (5)
Tremor (Nervous system disorders) | 10 (10) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 19 (19) | 23 (23)
Abdominal pain upper (Gastrointestinal disorders) | 24 (24) | 3 (3)
Constipation (Gastrointestinal disorders) | 35 (35) | 36 (36)
Diarrhea (Gastrointestinal disorders) | 65 (65) | 67 (67)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 29 (29) | 25 (25)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 16 (16) | 9 (9)
Gingival bleeding (Gastrointestinal disorders) | 6 (6) | 9 (9)
Hemorrhoids (Gastrointestinal disorders) | 10 (10) | 9 (9)
Mouth hemorrhage (Gastrointestinal disorders) | 12 (12) | 10 (10)
Nausea (Gastrointestinal disorders) | 85 (85) | 89 (89)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 7 (7)
Vomiting (Gastrointestinal disorders) | 57 (57) | 70 (70)
Hematuria (Renal and urinary disorders) | 10 (10) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 11 (11) | 14 (14)
Hair color changes (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
Petechiae (Skin and subcutaneous tissue disorders) | 32 (32) | 29 (29)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 22 (22) | 24 (24)
Skin lesion (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (19) | 17 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (16) | 10 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 14 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (17) | 22 (22)
Decreased appetite (Metabolism and nutrition disorders) | 46 (46) | 43 (43)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (13) | 11 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (15) | 18 (18)
Hypokalemia (Metabolism and nutrition disorders) | 27 (27) | 33 (33)
Hypomagnesemia (Metabolism and nutrition disorders) | 17 (17) | 19 (19)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7) | 9 (9)
Oral candidiasis (Infections and infestations) | 9 (9) | 10 (10)
Oral herpes (Infections and infestations) | 12 (12) | 9 (9)
Pneumonia (Infections and infestations) | 2 (2) | 15 (15)
Sinusitis (Infections and infestations) | 3 (3) | 9 (9)
Urinary tract infection (Infections and infestations) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No